CLINICAL TRIAL: NCT00264329
Title: Transitional Case Management Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Connecticut State, Department of Mental Health and Addiction Services (Other Government); National Development and Research Institutes, Inc. (Other); University of Delaware (Other); University of Kentucky (Other)
Responsible Party: Michael Prendergast/Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U01DA016211 (NIH)
Record Dates: First submitted 2005-12-08; First posted 2005-12-12 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Substance-Related Disorders
MeSH Terms: conditions — Substance-Related Disorders

INTERVENTIONS:
Other: Transitional Case Management Study — In an effort to address problems involved in parole re-entry, the Transitional Case Management (TCM) intervention tested a model of strengths-based case management consisting of (1) completion by the inmate of a strengths and goals assessment as part of discharge planning, (2) a telephone conference call that included the inmate and people central to the inmate's aftercare plan (including the parole officer), and (3) strengths case management for 12 weeks in the community to promote treatment participation and increase the client's access to needed services.

SUMMARY:
To address the issues involved in treatment participation by substance-abusing parolees, the CJ-DATS Transitional Case Management (TCM) study proposes to test a parole re-entry model that consists of (1) completion by the inmate of a strengths and goals assessment as part of discharge planning, (2) a telephone case conference call that includes the inmate and significant members of the inmate's aftercare plan (including the parole officer), and (3) strengths case management (for 12 weeks) in the community to promote treatment participation and support the client's access to needed services.

DETAILED DESCRIPTION:
To address the issues involved in treatment participation by substance-abusing parolees, the CJ-DATS Transitional Case Management (TCM) study proposes to test a parole re-entry model that consists of (1) completion by the inmate of a strengths and goals assessment as part of discharge planning, (2) a telephone case conference call that includes the inmate and significant members of the inmate's aftercare plan (including the parole officer), and (3) strengths case management (for 12 weeks) in the community to promote treatment participation and support the client's access to needed services.

More specifically, the multi-site study will evaluate the effects of a strengths case-management intervention on community-based treatment/service admission, retention, and utilization among inmates released from supervised treatment programs. If the intervention is successful, its wider adoption would increase the likelihood that inmates enter and remain in community services.

The specific aims of this multi-site study are to:

1. Increase the likelihood that offenders leaving prison (or other supervised setting) with a referral to community aftercare program services enroll in treatment.
2. Increase the amount of time that such offenders participate in community treatment.
3. Assist clients to get the services that they need during the first 12 weeks of return to the community.
4. As a result of the above, reduce relapse and reoffending during and following treatment.
5. Achieve the above results at a favorable cost-effectiveness ratio.
6. Encourage closer collaboration between the treatment and criminal justice systems.

Study participants (200 at each site, 25% of will be women) will be recruited in prison (or other confined setting) from inmates who have a referral to community treatment. After informed consent and a baseline interview, they will be randomly assigned to one of two conditions: (1) the Transitional Case Management condition, and (2) the Standard Referral condition (i.e., usual transition/re-entry procedures used by the facility, including a referral to community treatment).

Individual-level outcomes will include (1) treatment admission and participation (based on data collected from programs), (2) drug use, criminal activity, and psychosocial functioning (based on telephone interviews conducted 3 months after the end of the intervention) and (3) recidivism (based on records collected 12 months after the end of the intervention). The study will also assess the impact of the intervention on organizational and system factors (based on information from the case manager, treatment staff, and criminal justice staff) and the cost effectiveness of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Participate in a treatment program within a correctional institution (prison, work release, community correctional facility)
* Have a referral to a community-based substance abuse treatment program (as arranged by correctional staff or treatment staff)
* Within about 3 months until release
* Being released to the metropolitan area where case manager activities are being conducted

Exclusion Criteria:

* Referral to formal case management services in the community (e.g., for offenders with co-occurring disorders)
* Inability to provide informed consent (as determined by a set of questions about the consent process)
* Registered sex offender (as determined by the institution)
* Parole requirements that would prevent participation in the study (e.g., INS hold for deportation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 812 (Actual)
Dates: Start 2004-11; Primary Completion 2006-04 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Treatment admission by three months following parole | Three months
Treatment retention by three months following parole | Three months
Drug use at nine months following parole | Nine months
Recidivism at nine months following parole | Nine months

SECONDARY OUTCOMES:
Education and employment at nine months following parole | Nine months
HIV risk behaviors at nine months following parole | Nine months

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Prendergast, Ph.D., Principal Investigator — University of California, Los Angeles; Jerome Cartier, M.S., Study Director — University of California, Los Angeles
Locations (4):
- United States (4):
  - University of California, Los Angeles, Los Angeles, California
  - Connecticut Department of Mental Health and Addiction Services, Hartford, Connecticut
  - University of Kentucky, Lexington, Kentucky
  - National Development and Research Institutes, Inc. (NDRI), New York, New York

REFERENCES:
- [Result] Prendergast M, Frisman L, Sacks JY, Staton-Tindall M, Greenwell L, Lin HJ, Cartier J. A multi-site, randomized study of strengths-based case management with substance-abusing parolees. J Exp Criminol. 2011 Sep;7(3):225-253. doi: 10.1007/s11292-011-9123-y. Epub 2011 Apr 21. PMID 21949490
- [Result] Prendergast M, Greenwell L, Cartier J, Sacks J, Frisman L, Rodis E, Havens JR. Adherence to Scheduled Sessions in a Randomized Field Trial of Case Management: The Criminal Justice-Drug Abuse Treatment Studies Transitional Case Management Study. J Exp Criminol. 2009 Sep;5(3):273-297. doi: 10.1007/s11292-009-9077-5. Epub 2009 Jul 4. PMID 20157623